CLINICAL TRIAL: NCT04201262
Title: A Phase 3, External Placebo-Controlled, Open-Label, Multicenter Study to Evaluate the Efficacy and Safety of Ravulizumab in Adult Patients With Neuromyelitis Optica Spectrum Disorder (NMOSD)
Brief Title: An Efficacy and Safety Study of Ravulizumab in Adult Participants With NMOSD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALXN1210-NMO-307; CHAMPION-NMO-307 (Other: Alexion Pharmaceuticals); 2019-003352-37 (EudraCT Number)
Record Dates: First submitted 2019-12-11; First posted 2019-12-17 (Actual); Results first posted 2023-08-09 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Neuromyelitis Optica; Neuromyelitis Optica Spectrum Disorder
Keywords: Neuromyelitis Optica; Neuromyelitis Optica Spectrum Disorder; Devic's Disease; Transverse Myelitis; Optic Neuritis; Relapse; Ravulizumab; Ultomiris; ALXN1210; CNS Autoimmune Disorders; Demyelinating Disorders; NMO; NMOSD
MeSH Terms: conditions — Neuromyelitis Optica; Myelitis, Transverse; Optic Neuritis; Recurrence; Demyelinating Diseases | interventions — ravulizumab

STUDY DESIGN:
Intervention Model Description: External Placebo-Controlled, Open-Label Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ravulizumab (Experimental): During the Primary Treatment Period, all participants will receive open-label ravulizumab via intravenous (IV) infusion starting on Day 1. The end of the Primary Treatment Period will be triggered when the last enrolled participant completes between 26 and 50 weeks in the study (depending on the number of adjudicated On-Trial Relapse observed).
  After completion of the Primary Treatment Period, all participants will have the opportunity to continue receiving ravulizumab in the Long-Term Extension Period of the study. For each participant, the Long-Term Extension Period continues for up to 3 years, or until ravulizumab is approved and/or available (in accordance with country-specific regulations), whichever occurs first.
  Interventions: Biological: Ravulizumab

INTERVENTIONS:
Biological: Ravulizumab — Participants will receive a weight-based loading dose of ravulizumab via IV infusion on Day 1, followed by weight-based maintenance doses on Day 15, then once every 8 weeks until end of the Long-Term Extension Period.
  Other Names: ALXN1210; Ultomiris

SUMMARY:
The primary purpose of this study is to evaluate the efficacy and safety of ravulizumab for the treatment of adult participants with NMOSD.

ELIGIBILITY:
Inclusion Criteria:

1. Anti-aquaporin-4 antibody-positive and a diagnosis of NMOSD as defined by the 2015 international consensus diagnostic criteria.
2. At least 1 attack or relapse in the last 12 months prior to the Screening Period.
3. Expanded Disability Status Scale score ≤7.
4. Participants who enter the study receiving supportive immunosuppressive therapy must be on a stable dosing regimen of adequate duration prior to Screening.
5. Body weight ≥40 kilograms.
6. Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

1. History of Neisseria meningitidis infection.
2. Human immunodeficiency virus (HIV) infection (evidenced by HIV-1 or HIV-2 antibody titer).
3. Previously or currently treated with a complement inhibitor.
4. Use of rituximab or mitoxantrone within 3 months prior to Screening.
5. Use of IV immunoglobulin within 3 weeks prior to Screening.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (37):
- United States (10):
  - Research Site, Aurora, Colorado
  - Research Site, Fort Collins, Colorado
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Miami, Florida
  - Research Site, Boston, Massachusetts
  - Research Site, Rochester, Minnesota
  - Research Site, Jackson, Mississippi
  - Research Site, St Louis, Missouri
  - Research Site, Cincinnati, Ohio
  - Research Site, Houston, Texas
- Australia (2):
  - Research Site, Camperdown
  - Research Site, Fitzroy
- Research Site, Vienna, Austria
- Research Site, Burnaby, British Columbia, Canada
- Research Site, Aarhus, Denmark
- Research Site, Strasbourg, France
- Germany (3):
  - Research Site, Berlin
  - Research Site, Leipzig
  - Research Site, München
- Italy (5):
  - Research Site, Cefalù
  - Research Site, Gallarate
  - Research Site, Napoli
  - Research Site, Roma
  - Research Site, Rome
- Japan (5):
  - Research Site, Chiba
  - Research Site, Fukuoka
  - Research Site, Kawagoe-shi
  - Research Site, Niigata
  - Research Site, Sendai
- Poland (2):
  - Research Site, Katowice
  - Research Site, Lódz
- South Korea (2):
  - Research Site, Goyang-si
  - Research Site, Seoul
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Málaga
- Research Site, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Ortiz S, Pittock SJ, Berthele A, Levy M, Nakashima I, Oreja-Guevara C, Allen K, Mashhoon Y, Parks B, Kim HJ. Immediate and sustained terminal complement inhibition with ravulizumab in patients with anti-aquaporin-4 antibody-positive neuromyelitis optica spectrum disorder. Front Neurol. 2024 Jan 31;15:1332890. doi: 10.3389/fneur.2024.1332890. eCollection 2024. PMID 38356884
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ALXN1210-NMO-307&attachmentIdentifier=2dbb5864-d9d7-40e0-8e73-178d8adad5e4&fileName=ALXN1210-NMO-307_CSR_Synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study utilized the placebo group from Study ECU-NMO-301 (NCT01892345) as an external placebo control.
Groups:
- Ravulizumab: Participants received a weight-based loading dose of ravulizumab via intravenous (IV) infusion on Day 1, followed by weight-based maintenance doses on Day 15, then once every 8 weeks until the end of primary treatment period (up to 2.25 years). After the primary treatment period, participants continued to receive ravulizumab during the Long-Term Extension Period for up to approximately 2.63 years.
- Placebo (ECU-NMO-301): Participants who received eculizumab matching placebo in study ECU-NMO-301.
Period: Primary Treatment Period
Arm/Group | Ravulizumab | Placebo (ECU-NMO-301)
Started | 58 | 47
Received at Least 1 Dose of Study Drug | 58 | 47
Completed | 56 | 44
Not Completed | 2 | 3
Not completed — Adverse Event | 1 | 2
Not completed — Physician Decision | 1 | 1
Period: Long-term Extension Period
Arm/Group | Ravulizumab | Placebo (ECU-NMO-301)
Started | 56 | 0 (This arm was a placebo group from Study ECU-NMO-301 (an external placebo control). No participants from Study ECU-NMO-301 were enrolled into the long-term extension period in study ALXN1210-NMO-307.)
Received at Least 1 Dose of Study Drug | 56 | 0
Completed | 55 | 0
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety set included all participants who received at least 1 dose of study drug (ravulizumab or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Ravulizumab | Placebo (ECU-NMO-301) | Total
Number analyzed (Participants) | 58 | 47 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 44 | 95
  >=65 years | 7 | 3 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 42 | 94
  Male | 6 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 3 | 12
  Not Hispanic or Latino | 45 | 41 | 86
  Unknown or Not Reported | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 21 | 15 | 36
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 8 | 14
  White | 29 | 24 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Adjudicated On-trial Relapse in the Primary Treatment Period
Description: An On-trial Relapse was defined as a new onset of neurologic symptoms or worsening of existing neurologic symptoms with an objective change (clinical sign) on neurologic examination that persisted for more than 24 hours as confirmed by the treating physician. An adjudicated On-trial Relapse was defined by the protocol and positively adjudicated by the independent relapse adjudication committee.
Time Frame: Baseline up to 2.25 years (end of the Primary Treatment Period)
Population: The full analysis set (FAS) included all participants who had received at least 1 dose of study drug (ravulizumab or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Ravulizumab | Placebo (ECU-NMO-301)
Number analyzed (Participants) | 58 | 47
Participants | 0 | 20
Statistical Analysis 1: Comparison: Ravulizumab vs Placebo (ECU-NMO-301); Test type: Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.014, 95% CI 2-sided [0.000 to 0.103] — HR based on a Cox proportional hazards model, with Firth's adjustment. Confidence interval (CI)= Wald CI or Profile Likelihood CI Limits. HR for ravulizumab compared with placebo presented a 98.6% reduction in risk of relapse, 95% CI (89.7%, 100.0%)

2. Secondary Outcome: Adjudicated On-trial Annualized Relapse Rate (ARR) in the Primary Treatment Period
Description: The adjudicated On-trial ARR was computed as the total number of relapses divided by the total number of participant years in the study period. A central independent committee was used to adjudicate all On-trial Relapses as determined by the treating physician. Results reported as adjusted adjudicated On-trial ARR based on a Poisson regression centered on the mean historical ARR in the 24 months prior to screening.
Time Frame: Baseline up to 2.25 years (end of the Primary Treatment Period)
Population: The FAS included all participants who had received at least 1 dose of study drug (ravulizumab or placebo).
Measure: Number (95% Confidence Interval); unit: relapses/year on study
Arm/Group | Ravulizumab | Placebo (ECU-NMO-301)
Number analyzed (Participants) | 58 | 47
relapses/year on study | 0.000 [NA to NA] — Since there were no relapses, data could not be estimated. | 0.350 [0.199 to 0.616]

3. Secondary Outcome: Number of Participants With Clinically Important Change From Baseline in Hauser Ambulation Index (HAI) Score at the End of Primary Treatment Period
Description: The HAI is a rating scale developed to assess mobility by evaluating the time and degree of assistance required to walk 25 feet. The scale ranges from 0 to 9, with 0 being the best score (asymptomatic; fully ambulatory with no assistance) and 9 being the worst (restricted to wheelchair; unable to transfer self independently). Clinically important change is conditional on the baseline value: worsening if the baseline HAI is 0 and at least 2 points increase or if the baseline HAI is >0 and at least 1 point increase; improvement if the baseline value is at least 2 and at least 1 point decrease; and stable if baseline is 0 or 1 and a 0- or 1-point increase or decrease or baseline is at least 2 and not change.
Time Frame: Baseline up to 2.25 years (end of the Primary Treatment Period)
Population: The FAS included all participants who had received at least 1 dose of study drug (ravulizumab or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Ravulizumab | Placebo (ECU-NMO-301)
Number analyzed (Participants) | 58 | 47
Participants
  Clinical Improvement | 4 | 4
  Stable | 52 | 32
  Clinical Worsening | 2 | 11
Statistical Analysis 1: Comparison: Ravulizumab vs Placebo (ECU-NMO-301); The test of proportional odds was determined from a score test. The proportional odds was evaluated in univariate models; Test type: Other; p = 0.0122, Univariate models — Proportional Odds p-value

4. Secondary Outcome: Change From Baseline in European Quality of Life Health 5-dimension Questionnaire (EQ-5D) Index Score at the End of Primary Treatment Period
Description: The EQ-5D is a generic, standardized, self-administered instrument that provides a simple, descriptive profile and a single index value for health status. It consists of 2 parts; the EQ-5D descriptive system and the EQ-5D visual analogue scale (VAS). The EQ-5D descriptive system includes 5 dimensions; mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension measured on 3 levels: "no problem" (level 1), "some problems" (level 2), "extreme problems" (level 3). The digits for 5 dimensions can be combined in a 5-digit number describing the respondent's health state. The 5 dimensional 3-level systems was converted into single index utility score that ranges from less than 0 to 1, with higher scores representing a better health status.
Time Frame: Baseline, up to 2.25 years (end of the Primary Treatment Period)
Population: The FAS included all participants who had received at least 1 dose of study drug (ravulizumab or placebo).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ravulizumab | Placebo (ECU-NMO-301)
Number analyzed (Participants) | 58 | 47
units on a scale | 0.005 (0.1522) | -0.043 (0.2115)

5. Secondary Outcome: Change From Baseline in EQ-5D Visual Analog Scale (VAS) Score at the End of Primary Treatment Period
Description: The EQ-5D is a generic, standardized, self-administered instrument that provides a simple, descriptive profile and a single index value for health status. It consists of 2 parts; the EQ-5D descriptive system and the EQ-5D visual analogue scale (VAS). The EQ-5D VAS is an overall health state scale where the participant selects a number between 0 to 100 to describe the condition of their health, with 100 being 'The best health state you can imagine' and 0 being 'The worst health state you can imagine'. An increase in score indicates improvement.
Time Frame: Baseline, up to 2.25 years (end of the Primary Treatment Period)
Population: The FAS included all participants who had received at least 1 dose of study drug (ravulizumab or placebo).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ravulizumab | Placebo (ECU-NMO-301)
Number analyzed (Participants) | 58 | 47
units on a scale | 2.6 (14.07) | 0.6 (16.39)

6. Secondary Outcome: Number of Participants With Clinically Important Worsening From Baseline in Expanded Disability Status Scale (EDSS) Score at the End of Primary Treatment Period
Description: Disease-related disability was measured by the EDSS. The EDSS is an ordinal clinical rating scale that ranges from 0 (normal neurologic examination) to 10 (death) in half-point increments. Clinically important worsening was defined as an increase in EDSS score conditional on the baseline value: If the baseline EDSS was 0 and at least 2-point increase; if the baseline is 1 to 5, and at least 1-point increase; if the baseline is > 5 and at least 0.5 increase.
Time Frame: Baseline up to 2.25 years (end of the Primary Treatment Period)
Population: The FAS included all participants who had received at least 1 dose of study drug (ravulizumab or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Ravulizumab | Placebo (ECU-NMO-301)
Number analyzed (Participants) | 58 | 47
Participants
  No clinically important worsening | 52 | 36
  Clinically important worsening | 6 | 11

7. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Treatment-emergent Serious Adverse Events (TESAEs), and TEAEs Leading to Study Drug Discontinuation in the Primary Treatment Period
Description: An AE was as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An SAE was an AE that met at least 1 of the following criteria: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization for the AE, persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug), important medical event or reaction. TEAEs were AEs with a start date on or after the date of the first dose of study drug. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Baseline up to 2.25 years (end of the Primary Treatment Period)
Population: The safety set included all participants who received at least 1 dose of study drug (ravulizumab or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Ravulizumab | Placebo (ECU-NMO-301)
Number analyzed (Participants) | 58 | 47
Participants
  Any TEAEs | 53 | 45
  TESAEs | 8 | 26
  TEAEs Leading to Study Drug Discontinuation | 1 | 2

8. Secondary Outcome: Serum Ravulizumab Concentration
Time Frame: Predose and end of infusion (EOI) at Week 26
Population: Pharmacokinetics/pharmacodynamics (PK/PD) analysis set included participants who received at least 1 dose of study drug and who had at least 1 evaluable PK or PD result. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: micrograms (µg)/milliliter (mL)
Arm/Group | Ravulizumab
Number analyzed (Participants) | 56
micrograms (µg)/milliliter (mL)
  Week 26: Predose: number analyzed (Participants) | 55
  Week 26: Predose | 760.3 (202.75)
  Week 26: EOI | 1836.4 (355.39)

9. Secondary Outcome: Change From Baseline in Serum Free C5 Concentration at Week 26
Time Frame: Baseline, Week 26 (Predose and EOI)
Population: The PK/PD analysis set included participants who received at least 1 dose of study drug and who had at least 1 evaluable PK or PD result. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Ravulizumab
Number analyzed (Participants) | 55
µg/mL
  Change at Week 26: Predose: number analyzed (Participants) | 54
  Change at Week 26: Predose | -119.02 (42.857)
  Change at Week 26: EOI | -119.32 (42.512)

10. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADAs) During the Primary Treatment Period
Time Frame: Baseline, Weeks 26, 50, 82, and 106
Population: The safety set included all participants who received at least 1 dose of study drug (ravulizumab or placebo). Here, 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Ravulizumab
Number analyzed (Participants) | 58
Participants
  Baseline: Positive | 5
  Baseline: Negative | 53
  Week 26: number analyzed (Participants) | 55
  Week 26: Positive | 1
  Week 26: Negative | 54
  Week 50: number analyzed (Participants) | 52
  Week 50: Positive | 0
  Week 50: Negative | 52
  Week 82: number analyzed (Participants) | 15
  Week 82: Positive | 0
  Week 82: Negative | 15
  Week 106: number analyzed (Participants) | 1
  Week 106: Positive | 0
  Week 106: Negative | 1

ADVERSE EVENTS:
Time Frame: Up to approximately 4.9 years.
Description: The safety set included all participants who received at least 1 dose of study drug (ravulizumab or placebo). Per pre-specified analysis, data for the placebo arm (study ECU-NMO-301) was specified to be reported for primary analysis results only. Data were collected and are reported for the ravulizumab arm for the primary treatment period and long-term extension period separately.
Groups:
- Primary Treatment Period: Placebo: Participants who received eculizumab matching placebo in study ECU-NMO-301.
- Primary Treatment Period: Ravulizumab; Long-Term Extension: Ravulizumab: Participants received a weight-based loading dose of ravulizumab via intravenous (IV) infusion on Day 1, followed by weight-based maintenance doses on Day 15, then once every 8 weeks until the end of primary treatment period (up to 2.25 years). After the primary treatment period, participants continued to receive ravulizumab during the Long-Term Extension Period for up to approximately 2.63 years.
Arm/Group | Primary Treatment Period: Placebo | Primary Treatment Period: Ravulizumab | Long-Term Extension: Ravulizumab
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/58 | 1/56
Serious Adverse Events (participants affected / at risk) | 26/47 | 8/58 | 9/56
Other Adverse Events (participants affected / at risk) | 43/47 | 53/58 | 49/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Primary Treatment Period: Placebo (N=47) | Primary Treatment Period: Ravulizumab (N=58) | Long-Term Extension: Ravulizumab (N=56)
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Encephalitis meningococcal (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 0
Intervertebral discitis (Infections and infestations) | 0 | 1 | 0
Meningococcal sepsis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Pneumococcal infection (Infections and infestations) | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Myelitis transverse (Nervous system disorders) | 1 | 0 | 0
Neuromyelitis optica spectrum disorder (Nervous system disorders) | 16 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neuromyelitis optica pseudo relapse (Nervous system disorders) | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Treatment Period: Placebo (N=47) | Primary Treatment Period: Ravulizumab (N=58) | Long-Term Extension: Ravulizumab (N=56)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (2) | 3 (3) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 3 (3) | 3 (3)
Ear pain (Ear and labyrinth disorders) | 2 (3) | 1 (1) | 0 (0)
Paraesthesia ear (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Thyroid cyst (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
Blepharitis (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Eye disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Ocular discomfort (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal degeneration (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 4 (5) | 0 (0)
Vomiting (Gastrointestinal disorders) | 8 (10) | 4 (5) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 6 (14) | 3 (3) | 5 (6)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (5) | 3 (4) | 1 (1)
Nausea (Gastrointestinal disorders) | 12 (17) | 2 (2) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Alveolar bone resorption (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 1 (2) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 1 (3) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Angular cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Colitis microscopic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lip blister (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lip pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Presbyoesophagus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Allergy to arthropod bite (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 2 (2) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 14 (15) | 16 (16)
Urinary tract infection (Infections and infestations) | 9 (12) | 6 (7) | 6 (14)
Cystitis (Infections and infestations) | 1 (1) | 5 (7) | 2 (3)
Upper respiratory tract infection (Infections and infestations) | 6 (10) | 5 (5) | 6 (12)
Nasopharyngitis (Infections and infestations) | 8 (12) | 3 (3) | 4 (6)
Sinusitis (Infections and infestations) | 0 (0) | 3 (3) | 2 (2)
Conjunctivitis (Infections and infestations) | 4 (8) | 2 (2) | 0 (0)
Oral herpes (Infections and infestations) | 2 (2) | 3 (3) | 4 (6)
Periodontitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasal herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Post-acute COVID-19 syndrome (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Stenotrophomonas infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tinea versicolour (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Viral pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Body tinea (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Chronic tonsillitis (Infections and infestations) | 1 (3) | 0 (0) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mastitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 3 (6) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (3) | 1 (1) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Chillblains (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (6) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 4 (8) | 0 (0) | 1 (2)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (3) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Post procedural contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 2 (2) | 1 (1) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 1 (1) | 1 (1)
Urinary occult blood (Investigations) | 0 (0) | 1 (2) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood pressure systolic increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Bone density decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Cortisol decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 1 (2) | 0 (0) | 0 (0)
Gardnerella test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 3 (3) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Folate deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (9) | 7 (8) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (9) | 6 (6) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (11) | 2 (2) | 2 (3)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pelvic deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Fracture pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Synovial disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 10 (17) | 15 (25) | 5 (6)
Dizziness (Nervous system disorders) | 6 (6) | 4 (4) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 3 (4) | 0 (0)
Paraesthesia (Nervous system disorders) | 3 (4) | 2 (3) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 4 (5) | 1 (1) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0)
Parosmia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sensory disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Head discomfort (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Mental impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle contractions involuntary (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasticity (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Uhthoff's phenomenon (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 2 (2) | 2 (2)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 4 (5) | 1 (1) | 3 (3)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep talking (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Delusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Obsessive-compulsive disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Persistent depressive disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 2 (3) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Strangury (Renal and urinary disorders) | 0 (0) | 1 (5) | 1 (1)
Cystitis interstitial (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Glycosuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Prerenal failure (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Urethral syndrome (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Menopausal symptoms (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 3 (3) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tonsillolith (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (8) | 1 (1) | 2 (2)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Sensitive skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Menopause (Social circumstances) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 2 (2) | 1 (2)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (3) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Macrocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Heart failure with preserved ejection fraction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eyelid ptosis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal fat apron (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatic cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Bacterial vulvovaginitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Coronavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Immunisation reaction (Injury, poisoning and procedural complications) | 1 (1) | 2 (3) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural headache (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Antinuclear antibody positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Culture cervix positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Protein urine present (Investigations) | 0 (0) | 0 (0) | 1 (1)
Red blood cell sedimentation rate increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 1 (2)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Temporomandibular pain and dysfunction syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Benign soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Migraine with aura (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neuromyelitis optica pseudo relapse (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Partial seizures with secondary generalisation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Cystitis-like symptom (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Cough variant asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Paranasal sinus inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural thickening (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Androgenetic alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Anorectal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 2 (2) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 2 (2) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (12) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 3 (5) | 0 (0)
Cyst (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 5 (5) | 3 (3) | 1 (1)
Feeling cold (General disorders) | 1 (2) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Induration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (3) | 1 (2) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 3 (3) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 0 (0) | 1 (1)
Pain (General disorders) | 4 (7) | 2 (2) | 0 (0)
Peripheral swelling (General disorders) | 2 (3) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 4 (5) | 5 (6) | 1 (1)
Swelling face (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vaccination site pain (General disorders) | 0 (0) | 3 (3) | 1 (1)
Vaccination site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Otitis media chronic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Foreign body (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Spinal retrolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Medical device entrapment (Product Issues) | 0 (0) | 0 (0) | 1 (1)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Lactation insufficiency (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT04201262/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-25): https://cdn.clinicaltrials.gov/large-docs/62/NCT04201262/SAP_002.pdf